CLINICAL TRIAL: NCT04468880
Title: Effect of Milk Consumption, Containing A2 β-caseins Only, on Digestive Comfort. A Randomized and Double-blind Study
Brief Title: Milk Consumption on Digestive Comfort.
Acronym: A2-DIGEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD in nutrition and endocrinology, Institut Pasteur de Lille
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2020-A00185-34
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: milk intolerant; β-caseins A1 and A2; Lactose
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: monocentric, double-blind, randomized, controlled, cross-over and ambulatory study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk A1A2 (Other): Group (A1 → A2) receiving control milk A1A2 in period 1 then the milk evaluated A2A2 in period 2
  Interventions: Other: Group (A1 → A2)
- Milk A2A2 (Other): Group (A2 → A1) receiving the milk evaluated A2A2 in period 1 then the control milk A1A2 in period 2
  Interventions: Other: Group (A2 → A1)

INTERVENTIONS:
Other: Group (A1 → A2) — Before each start of consumption of the products under study, a wash-out period of 2 weeks (no consumption of milk) must be observed by the subjects.
  25 subjects will consume A1A2 milk for 2 weeks (period 1), then they will consume A2A2 milk for 2 weeks (period 2).
  During each consumption period, various questionnaires will be completed by the subjects: frequency and consistency of stool, analog visual scales on digestive comfort and dietary surveys. Stool collections will also be carried out.
  Arms: Milk A1A2
Other: Group (A2 → A1) — Before each start of consumption of the products under study, a wash-out period of 2 weeks (no consumption of milk) must be observed by the subjects.
  25 subjects will consume A2A2 milk for 2 weeks (period 1), then they will consume A1A2 milk for 2 weeks (period 2).
  During each consumption period, various questionnaires will be completed by the subjects: frequency and consistency of stool, analog visual scales on digestive comfort and dietary surveys. Stool collections will also be carried out.
  Arms: Milk A2A2

SUMMARY:
Lactose, naturally present in milk, can cause digestive discomfort. Delactosed milk is currently the only one alternative to cow's milk for intolerant people. As some of them do not digest milk, it was completely remove from their diet. However, are they really intolerant to lactose or intolerant to milk (or to another of its compounds)? Do β-caseins play a role in this intolerance? β-caseins are proteins naturally present in milk. Two types of β-caseins were identified: A1 and A2. These types differ according to the genetic profile of the cow and depend on the breed. The rare clinical studies interested in this topic suggest that:

1. consumption of milk A1 versus consumption of milk A2 can lead to: softer stools, delayed transit, as well as pro-inflammatory effects in some individuals,
2. consumption of A2 milk significantly reduces gastrointestinal symptoms and improves digestive comfort in lactose intolerant people.

Thus, it would be interesting to be able to assess the effect of a consumption of A2A2 milk type compared to A1A2 milk type, both on the parameters of digestive comfort and on inflammatory parameters.

DETAILED DESCRIPTION:
The study will be carried out on healthy volunteers, aged 18 to 65 and self-declared sensitive, even intolerant to the consumption of milk.

The main objective of the study is to assess the impact of milk β-caseins (A2A2 vs A1A2) on the digestive comfort felt during the consumption of milk in subjects declaring that they do not tolerate milk.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman;
* 18 to 65 years old;
* Declaring to have sensitivity or intolerance when consuming cow's milk;
* Agreeing to follow the constraints generated by the study;
* Having signed the informed consent form;
* Social insured.

Exclusion Criteria:

* Subject with an allergy to cow's milk proteins;
* Subject suffering from a severe eating disorder (anorexia, bulimia, binge eating);
* Subject with chronic pathology interfering with the parameters studied during this study (inflammatory intestinal disease, celiac disease);
* Subject suffering from acute intestinal infection at the time of inclusion (gastroenteritis, etc.);
* Subject with immunodeficiency or any other serious pathology (cancer, hemopathy);
* Pregnant or planning to be pregnant during the study period;
* Subject participating in another clinical study or in period of exclusion from another study;
* Subject deprived of liberty;
* Subject under judicial protection measure;
* Whose main investigator or a qualified co-investigator judges that the state of health or the concomitant treatments are not compatible with the good progress of the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Analog visual scales | 4 weeks
  Digestive comfort will be assessed daily by the average of the following analog visual scales (score : 0 to 10), completed within 30 min to 3 hours after consumption of the daily dose of milk, depending on the usual occurrence of symptoms in individuals:
  * I have bloating
  * I have abdominal pain
  * I have flatulence (gas)
  * I have borborygmas (gurgling)
  * I have reflux (return, rise)
  * Overall, I estimate my digestive comfort.
  The average of these 6 analog visual scales, called Global Digestive Discomfort (IDG), will therefore be available every day for 14 days; the final variable analyzed will be the average of these 14 IDG values, and will be called Global Average Digestive Discomfort (IDGM).

SECONDARY OUTCOMES:
Analysis of the average per period of each analog visual scales independently | 4 weeks
  The analogue visual scales will be completed daily during each period of milk consumption (4 weeks)
Difference Calprotectin at the end of the period - Calprotectin at V0 (measured in mg/kg) | 4 weeks
  Stool collections are made during inclusion visits, V1 follow-up and V3 end of study.
For each of the inflammatory markers (CRP us, IL-1β, TNF-α, IL-6) : difference between value at the end of the period and value at V0 | 4 weeks
  Blood samples are taken during inclusion visits, V1 follow-up and V3 end of study.
  All of the inflammatory markers are measured in pg/ml.
Average stool frequencies and consistencies | 4 weeks
  This questionnaires will be completed daily during each period of milk consumption (4 weeks).
  Bristol scale: stool type 1 (separate hard balls) to stool type 7 (watery, structureless stools)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: Undecided